CLINICAL TRIAL: NCT00084656
Title: An Extended Dosing, Two-phase Study of MDX-010 as Monotherapy or in Combination With Tyrosinase/gp100/MART-1 Peptides Emulsified With Montanide ISA 51 VG in the Treatment of Subjects With Resected Stage III or Stage IV Melanoma
Brief Title: Monoclonal Antibody Therapy and Vaccine Therapy in Treating Patients With Resected Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365467; P30CA076292 (NIH); P30CA014089 (NIH); MCC-15241 (Other: Moffitt Cancer Center); MDX010-16 (Other: Medarex); NCI-6446 (Other: National Cancer Institute); CA184-016 (Other: BMS)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; recurrent melanoma; recurrent intraocular melanoma; metastatic intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Ipilimumab; Monophenol Monooxygenase

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: ipilimumab; Biological: Tyrosinase/gp100/MART-1 Peptides

INTERVENTIONS:
Biological: ipilimumab — IV over 90 mins on day 1, wks 1,9,17,25,33,41,53 Dose: 3 mg/kg (Part I), 10 mg/kg (Part II)
Biological: Tyrosinase/gp100/MART-1 Peptides — (All subjects in Part I and HLA-A*0201 positive subjects only in Part II): SC, day 1 of wks 1,3,5,7,9,11,17, 21,25,33,41,53 Dose: 1 mg peptide emulsified in 1 mL Montanide ISA 51 VG.)

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Vaccines may make the body build an immune response to kill tumor cells. Combining the vaccines with Montanide ISA-51 may cause a stronger immune response and kill more tumor cells. Giving monoclonal antibody therapy together with vaccine therapy may be an effective treatment for stage III or stage IV melanoma.

PURPOSE: This phase II trial is studying how well giving monoclonal antibody therapy together with vaccine therapy works in treating patients with resected stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Achieve at least a 40% autoimmune breakthrough event rate, as defined by the induction of grade 1, grade 2, or acceptable grade 3 drug-related autoimmune adverse events, in patients with resected stage III or IV melanoma treated with anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen emulsified in Montanide ISA-51.

Secondary

* Determine the incidence of drug-related autoimmune adverse events of any grade in patients treated with this regimen.
* Determine the time to disease relapse in patients treated with this regimen.
* Determine the immunologic response in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) IV over 90 minutes on day 1 of weeks 1, 9, 17, 25, 33, 41, and 53 and peptide vaccine comprising tyrosinase, gp100 antigen, and MART-1 antigen emulsified in Montanide ISA-51 subcutaneously on day 1 of weeks 1, 3, 5, 7, 9, 11, 17, 21, 25, 33, 41, and 53.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Stage III (≥ 3 positive lymph nodes) or stage IV disease
  * Mucosal or ocular melanoma allowed
* Completely resected within the past 6 months
* Patients with stage III resected melanoma rendered free of disease may have failed, been ineligible for, or refused prior treatment with interferon alfa
* Positive staining of tumor tissue for at least one of the following:

  * Antibody HMB-45 for gp100
  * Antibody HMB-45 for tyrosinase
  * Antibody HMB-45 for MART-1
* HLA-A*0201 positive by DNA allele-specific polymerase chain reaction assay

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* WBC ≥ 2,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hematocrit ≥ 30%
* Hemoglobin ≥ 10 g/dL

Hepatic

* AST ≤ 3 times upper limit of normal (ULN)*
* Bilirubin ≤ ULN* (< 3.0 mg/dL for patients with Gilbert's syndrome)
* No significant hepatic disease that would preclude study participation
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative NOTE: * Unless attributable to disease

Renal

* Creatinine ≤ 2.0 mg/dL
* No significant renal disease that would preclude study participation

Cardiovascular

* No significant cardiac disease that would preclude study participation

Pulmonary

* No significant pulmonary disease that would preclude study participation

Immunologic

* No history of any of the following:

  * Inflammatory bowel disease or any other autoimmune bowel disease
  * Systemic lupus erythematosus
  * Rheumatoid arthritis
  * Autoimmune ocular disease
* No systemic hypersensitivity to Montanide ISA-51 or any vaccine component
* No active infection requiring therapy
* HIV negative

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No significant gastrointestinal disease that would preclude study participation
* No significant psychiatric disease that would preclude study participation
* No other medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010)
* No prior gp100 antigen, MART-1 antigen, or tyrosinase peptide
* At least 4 weeks since prior immunotherapy for melanoma and recovered
* No other concurrent immunotherapy

Chemotherapy

* At least 4 weeks since prior chemotherapy for melanoma (6 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy

Endocrine therapy

* At least 4 weeks since prior hormonal therapy for melanoma and recovered
* At least 4 weeks since prior systemic, inhaled, or topical corticosteroids
* No concurrent systemic, inhaled, or topical corticosteroids

Radiotherapy

* At least 4 weeks since prior radiotherapy for melanoma and recovered

Surgery

* See Disease Characteristics
* At least 4 weeks since prior surgery for melanoma and recovered

Other

* No concurrent immunosuppressive agents (e.g., cyclosporine and its analog)
* Concurrent analgesic therapy allowed provided the dose is stable for the past 14 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-05-31 (Actual); Primary Completion 2009-10-31 (Actual); Study Completion 2009-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Garg SK, Ott MJ, Mostofa AGM, Chen Z, Chen YA, Kroeger J, Cao B, Mailloux AW, Agrawal A, Schaible BJ, Sarnaik A, Weber JS, Berglund AE, Mule JJ, Markowitz J. Multi-Dimensional Flow Cytometry Analyses Reveal a Dichotomous Role for Nitric Oxide in Melanoma Patients Receiving Immunotherapy. Front Immunol. 2020 Feb 25;11:164. doi: 10.3389/fimmu.2020.00164. eCollection 2020. PMID 32161584
- [Derived] Sarnaik AA, Yu B, Yu D, Morelli D, Hall M, Bogle D, Yan L, Targan S, Solomon J, Nichol G, Yellin M, Weber JS. Extended dose ipilimumab with a peptide vaccine: immune correlates associated with clinical benefit in patients with resected high-risk stage IIIc/IV melanoma. Clin Cancer Res. 2011 Feb 15;17(4):896-906. doi: 10.1158/1078-0432.CCR-10-2463. Epub 2010 Nov 24. PMID 21106722

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 participants enrolled, 76 treated. 1 not treated due to protocol violation.
Groups:
- 3.0 MG/KG IPILIMUMAB + PEPTIDES: HLA-A*201 positive participants receive ipilimumab at 3 mg/kg/dose as an intravenous (i.v.) infusion every 8 weeks for 12 months for a total of 7 infusions.
  Peptides administered at Weeks 1, 3, 5, 7, 9, 11, 17, 21, 25, 33, 41, and 53 for a total of 12 vaccinations.
- 10 MG/KG IPILIMUMAB + PEPTIDES: HLA-A*201 positive participants receive ipilimumab at 10 mg/kg/dose as an intravenous (i.v.) infusion every 8 weeks for 12 months for a total of 7 infusions.
  Peptides administered at Weeks 1, 3, 5, 7, 9, 11, 17, 21, 25, 33, 41, and 53 for a total of 12 vaccinations.
- 10 MG/KG IPILIMUMAB: HLA-A*201 negative participants receive ipilimumab at 10 mg/kg/dose as an intravenous (i.v.) infusion every 8 weeks for 12 months for a total of 7 infusions.
Period: Overall Study
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Started | 25 | 25 | 26
Completed | 0 | 0 | 0
Not Completed | 25 | 25 | 26
Not completed — Other reasons | 0 | 12 | 11
Not completed — Withdrawal by Subject | 15 | 4 | 4
Not completed — Disease relapse | 0 | 9 | 10
Not completed — Disease progression | 9 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB | Total
Number analyzed (Participants) | 25 | 25 | 26 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (15.25) | 53.3 (10.34) | 51.5 (14.06) | 53.1 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 9 | 31
  Male | 13 | 15 | 17 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 1 | 1
  White | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immune-related Adverse Events (irAEs)
Description: Percentage of participants who experienced an irAE during the course of the study defined by the induction of Grade 1, Grade 2, or acceptable Grade 3 drug-related irAEs.
  For the purposes of this trial, acceptable drug-related irAEs are skin-related immune-mediated adverse events < or = Grade 3 (potentially reversible inflammation < Grade 4 that can be attributable to a local antitumor reaction that could potentially be a therapeutic response will also be considered an acceptable irAE).
  Note: The confidence interval was calculated using the Clopper Pearson method
Time Frame: Between first dose and 70 days after last dose of study therapy (up to 3 years including maintenance phase)
Population: All treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 25 | 25 | 26
Percentage of participants | 80.0 [62.5 to 91.8] | 72.0 [53.8 to 86.1] | 65.4 [47.4 to 80.6]

2. Primary Outcome: Time to Disease Relapse
Description: To determine the time (months) from first dose to disease relapse.
  Time to disease relapse is defined from the start of treatment to the first occurrence of any new lesion (reported by the investigator on physical exam or diagnostic imaging assessments that are attributed to metastatic melanoma) or death. Participants who neither relapse nor died will be censored on the date of their last tumor evaluation.
  Median estimated using Kaplan-Meier method; A two-sided 95% CI for median in each treatment group was computed via the log-log transformation method.
Time Frame: up to 3 years
Population: All treated participants for the 10 mg/kg ipilimumab arms of the study only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 25 | 26
Months | NA [10.38 to NA] — insufficient number of events to achieve median value determination and upper limit | NA [7.59 to NA] — insufficient number of events to achieve median value determination and upper limit

3. Secondary Outcome: Number of Participants With Drug-related irAEs of Any Grade
Description: The number of participants who experienced a drug-related irAE of any grade over the course of the study.
  Note: The confidence interval was calculated using the Clopper Pearson method
Time Frame: Between first dose and 70 days after last dose of study therapy (up to 3 years including maintenance phase)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 25 | 25 | 26
Participants | 24 | 24 | 24

4. Secondary Outcome: Immunologic Response to the Dose Regimen
Description: The secondary objective was to determine the immunologic response to the dosing regimen, via Human Anti-Human Antibody (HAHA) Assessment, displayed by number of participants observed as HAHA positive or negative.
  Note: If participant had at least one post-baseline HAHA result with increase in titer over pre-study, the participant is counted as HAHA Positive.
  A participant with all negative post-baseline results is counted as HAHA negative.
Time Frame: up to 3 years
Population: All Treated Subjects with Baseline and at Least one Post-Baseline HAHA Assessment
Measure: Number; unit: Number of participants
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 24 | 21 | 21
Number of participants
  HAHA positive at baseline | 5 | 1 | 0
  HAHA positive | 5 | 2 | 1
  HAHA negative | 19 | 19 | 20

5. Secondary Outcome: Number of Participants Experiencing Hematology-related Lab Abnormalities
Description: The number of participants who experienced a Hematology-related laboratory abnormality (grade 1-4 and grade 3-4 categories, grade 4 being the worst) during the course of the study.
  Laboratory tests were graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
Time Frame: Between first dose and 70 days after last dose of study therapy (up to 3 years including maintenance phase)
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 25 | 25 | 26
Number of participants
  White blood cells, grade 1-4 | 5 | 1 | 0
  White blood cells, grade 3-4 | 0 | 0 | 0
  Absolute Neutrophil Count, grade 1-4 | 6 | 2 | 3
  Absolute Neutrophil Count, grade 3-4 | 1 | 0 | 0
  Platelet Count, grade 1-4 | 4 | 2 | 1
  Platelet Count, grade 3-4 | 0 | 0 | 0
  Hemoglobin, grade 1-4 | 8 | 10 | 15
  Hemoglobin, grade 3-4 | 0 | 0 | 0
  Lymphocytes, grade 1-4 | 19 | 15 | 17
  Lymphocytes, grade 3-4 | 1 | 1 | 1

6. Secondary Outcome: Number of Participants Experiencing Serum Chemistry-related Lab Abnormalities
Description: The number of participants who experienced a Serum Chemistry-related laboratory abnormality (grade 1-4 and grade 3-4 categories, grade 4 being the worst) during the course of the study.
  Laboratory tests were graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
Time Frame: Between first dose and 70 days after last dose of study therapy (up to 3 years including maintenance phase)
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
Number analyzed (Participants) | 25 | 25 | 26
Number of participants
  alanine aminotransferase (ALT), grade 1-4: number analyzed (Participants) | 25 | 25 | 25
  alanine aminotransferase (ALT), grade 1-4 | 5 | 6 | 7
  alanine aminotransferase (ALT), grade 3-4: number analyzed (Participants) | 25 | 25 | 25
  alanine aminotransferase (ALT), grade 3-4 | 0 | 1 | 1
  aspartate aminotransferase (AST), grade 1-4: number analyzed (Participants) | 25 | 25 | 25
  aspartate aminotransferase (AST), grade 1-4 | 9 | 4 | 7
  aspartate aminotransferase (AST), grade 3-4: number analyzed (Participants) | 25 | 25 | 25
  aspartate aminotransferase (AST), grade 3-4 | 0 | 0 | 1
  Total Bilirubin, grade 1-4: number analyzed (Participants) | 25 | 25 | 25
  Total Bilirubin, grade 1-4 | 2 | 1 | 1
  Total Bilirubin, grade 3-4: number analyzed (Participants) | 25 | 25 | 25
  Total Bilirubin, grade 3-4 | 0 | 0 | 1
  Alkaline Phosphatase, grade 1-4: number analyzed (Participants) | 25 | 25 | 25
  Alkaline Phosphatase, grade 1-4 | 5 | 0 | 3
  Alkaline Phosphatase, grade 3-4: number analyzed (Participants) | 25 | 25 | 25
  Alkaline Phosphatase, grade 3-4 | 0 | 0 | 0
  Amylase, grade 1-4: number analyzed (Participants) | 18 | 25 | 26
  Amylase, grade 1-4 | 5 | 7 | 10
  Amylase, grade 3-4: number analyzed (Participants) | 18 | 25 | 26
  Amylase, grade 3-4 | 1 | 0 | 0
  Lipase, grade 1-4: number analyzed (Participants) | 18 | 25 | 26
  Lipase, grade 1-4 | 3 | 5 | 10
  Lipase, grade 3-4: number analyzed (Participants) | 18 | 25 | 26
  Lipase, grade 3-4 | 2 | 2 | 4
  Creatinine, grade 1-4 | 3 | 2 | 1
  Creatinine, grade 3-4 | 0 | 0 | 0

7. Secondary Outcome: Time to Disease Relapse
Description: as for outcome 2
Time Frame: up to 3 years
Population: All treated participants for the 3 mg/kg ipilimumab arm of the study only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES
Number analyzed (Participants) | 25
Months | NA [15.80 to NA] — insufficient number of events to achieve median value determination and upper limit

ADVERSE EVENTS:
Time Frame: From first dose to 70 days post last dose (up to 3 years)
Arm/Group | 3.0 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB + PEPTIDES | 10 MG/KG IPILIMUMAB
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 5/25 | 7/25 | 10/26
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3.0 MG/KG IPILIMUMAB + PEPTIDES (N=25) | 10 MG/KG IPILIMUMAB + PEPTIDES (N=25) | 10 MG/KG IPILIMUMAB (N=26)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 2 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Blood corticotrophin decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3.0 MG/KG IPILIMUMAB + PEPTIDES (N=25) | 10 MG/KG IPILIMUMAB + PEPTIDES (N=25) | 10 MG/KG IPILIMUMAB (N=26)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 1 | 3
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 3 | 4
Dry eye (Eye disorders) | 1 | 0 | 2
Eye pain (Eye disorders) | 1 | 2 | 0
Eye pruritus (Eye disorders) | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 1 | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2
Photophobia (Eye disorders) | 1 | 2 | 0
Vision blurred (Eye disorders) | 4 | 4 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 12 | 10
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 5 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 15 | 16 | 20
Flatulence (Gastrointestinal disorders) | 3 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 9 | 9 | 12
Vomiting (Gastrointestinal disorders) | 2 | 4 | 6
Chills (General disorders) | 8 | 6 | 8
Face oedema (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 24 | 19 | 20
Granuloma (General disorders) | 13 | 21 | 1
Influenza like illness (General disorders) | 14 | 7 | 2
Injection site erythema (General disorders) | 4 | 7 | 0
Injection site nodule (General disorders) | 14 | 1 | 0
Injection site pain (General disorders) | 17 | 13 | 0
Injection site pruritus (General disorders) | 8 | 5 | 0
Injection site rash (General disorders) | 5 | 1 | 0
Injection site reaction (General disorders) | 25 | 11 | 0
Injection site swelling (General disorders) | 2 | 3 | 0
Injection site vesicles (General disorders) | 2 | 0 | 0
Irritability (General disorders) | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 2 | 2
Oedema (General disorders) | 2 | 1 | 1
Oedema peripheral (General disorders) | 9 | 9 | 3
Pain (General disorders) | 3 | 1 | 2
Pyrexia (General disorders) | 12 | 10 | 8
Hypersensitivity (Immune system disorders) | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 6 | 2
Oral candidiasis (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2
Blood corticotrophin decreased (Investigations) | 0 | 0 | 3
Blood testosterone decreased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 4 | 3 | 7
Weight increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Amnesia (Nervous system disorders) | 1 | 3 | 0
Aphasia (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 5
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 8 | 13 | 14
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 2
Depression (Psychiatric disorders) | 3 | 1 | 3
Insomnia (Psychiatric disorders) | 4 | 3 | 6
Libido decreased (Psychiatric disorders) | 0 | 1 | 2
Sleep disorder (Psychiatric disorders) | 0 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 18 | 18
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 16 | 17 | 18
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 3 | 1 | 1
Varicose vein (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less